CLINICAL TRIAL: NCT05656924
Title: Improving the Health Status of Dysvascular Amputees by Deploying Digital Prosthetic Interface Technology in Combination With an Exercise Intervention
Brief Title: Deploying Digital Prosthetic Interface Technology and Exercise in Dysvascular Amputees
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: Bionic Skins LLC (Unknown); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Paolo Bonato, Director, Motion Analysis Laboratory, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022P003160; R44HD110327 (NIH)
Record Dates: First submitted 2022-12-08; First posted 2022-12-19 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Diabete Type 2; Amputation
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Study participants will be randomized to one of two groups: group 1 will use the digital prosthetic interface technology developed by Bionic Skins and group 2 will use a traditional socket-liner technology (i.e., study participants will use their own liner and socket system).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- digital prosthetic interface technology group (Experimental): Study participants randomized to this group will use the digital prosthetic interface technology developed by Bionic Skins.
  Interventions: Device: digital prosthetic interface technology
- traditional socket and liner technology group (No Intervention): Study participants randomized to this group will use a traditional socket-liner technology (i.e., study participants will use their own liner and socket system).

INTERVENTIONS:
Device: digital prosthetic interface technology — Individuals randomized to this group will receive a socket and liner that are manufactured using a novel technique meant to achieve a better distribution of pressure on the residuum. The study is based on the hypothesis that an improvement in pressure distribution on the residuum will enable high adherence to an exercise program meant to improve health status in dysvascular amputees.
  Arms: digital prosthetic interface technology group

SUMMARY:
The study will test a new approach to the design and implementation of socket and liner technology in individuals who lost a lower limb secondary to diabetes mellitus type II (herein referred to as dysvascular amputees). The technology-based intervention will be combined with an exercise program designed to improve the health status of dysvascular amputees.

DETAILED DESCRIPTION:
The study will test the hypothesis that the use of a digital approach to the design and implementation of socket and liner technology (herein referred to as "digital prosthetic interface technology") leads to better health of the residuum (compared to traditional socket and liner technology). This hypothesis will be tested by recruiting a group of dysvascular amputees (herein meant to refer to individuals who lost a lower limb secondary diabetes mellitus type II) and by randomizing them to either receiving a digital prosthetic interface technology or a traditional socket and liner system. Furthermore, the study will assess if the digital prosthetic interface technology improves adherence to an exercise program and results in better clinical outcomes. To test this hypothesis, an exercise intervention will be deployed by relying on coaching and mobile health technology to encourage adherence to a walking program targeting dysvascular transtibial amputees. This exercise intervention is an extension of pilot work that demonstrated the suitability of mobile health technology to implement an exercise-based intervention program in dysvascular amputees.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral transtibial amputation within the past 4-16 months
* Etiology secondary to complications of Diabetes Mellitus (DM) type II
* Current use of a prosthesis, with at least 2 months prior use
* K2 or K3 level (as determined using the Amputee Mobility Predictor assessment tool)
* Own a smartphone

Exclusion Criteria:

* Amputation due to cancer or macrotrauma or acute hemorrhage
* Bilateral amputation
* Medically or surgically unstable contralateral lower extremity as determined by medical criteria (e.g., critical limb ischemia)
* Severe residual limb pain that limits function preventing participation in an exercise-based program
* Medical conditions that would interfere with subject's participation in regular sustained exercise
* Anthropometric characteristics that are not compatible with the technology used to scan the residuum and manufacture the liner and socket (e.g., a residuum circumference greater than 32 inches would not be compatible with the device used to scan the residuum)
* Current pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in intra-socket interface pressure between the two groups | Baseline
  Pressure sensors inserted in the socket will be used to measure the pressure on the residuum when study participants are weight bearing. The pressure is measured in kilopascals (kPa). 1 kPa is approximately the pressure exerted by a 10-g mass resting on a 1-cm2 area.
Difference in step counts between the two groups | 12 months
  The average number of steps over a period of 2 weeks will be provided by a wearable sensor (Oura ring). The data will be expressed in number of steps per day.

SECONDARY OUTCOMES:
Difference in thermal imaging measures of the temperature of the residuum in the two groups | Baseline
  A thermal camera will be used to measure the peak temperature of the residuum. The residuum temperature will be measured in degrees Celsius.
Difference in Socket Evaluation Questionnaire (SEQ) scores in the two groups | Baseline
  The Socket Evaluation Questionnaire (SEQ) consists of a battery of questions inquiring about subject's comfort using a socket. The SEQ uses a visual analog scale format. The output ranges from 0 (worst) to 100 (best).
Difference in Prosthesis Evaluation Questionnaire (PEQ) scores in the two groups | Baseline
  The Prosthesis Evaluation Questionnaire (PEQ) consists of a battery of questions inquiring about subject's perception of his/her prosthesis. The PEQ uses a visual analog scale format. The output ranges from 0 (worst) to 100 (best).

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Bonato, PhD, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No